CLINICAL TRIAL: NCT03892980
Title: A Prospective, Multicenter Investigation of the da Vinci® Surgical Systems in Nipple Sparing Mastectomy (NSM) Procedures
Brief Title: Robotic-Assisted da Vinci System Prophylactic Nipple-Sparing Mastectomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ISI dV Xi-SP NSM
Record Dates: First submitted 2019-03-21; First posted 2019-03-27 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Nipple Sparing Mastectomy
Keywords: breast; robot; robotic; nipple sparing mastectomy; NSM; da Vinci; surgery; mastectomy; prophylactic NSM; risk reducing; BRCA mutation; nipple areola complex; NAC; RNSM; high-risk genetic mutation; gene mutation
MeSH Terms: interventions — Mastectomy, Subcutaneous

STUDY DESIGN:
Intervention Model Description: Subjects undergo nipple-sparing mastectomy (NSM) procedures using the da Vinci Surgical Systems
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Nipple Sparing Mastectomy (Experimental)
  Interventions: Device: Nipple-Sparing Mastectomy

INTERVENTIONS:
Device: Nipple-Sparing Mastectomy — Nipple-sparing mastectomy using da Vinci Surgical Systems.

SUMMARY:
This study evaluates the safety and effectiveness of the da Vinci Surgical Systems in prophylactic Nipple Sparing Mastectomy procedures.

DETAILED DESCRIPTION:
Surgical management for breast cancer and risk-reducing techniques have evolved from radical mastectomy to other techniques such as nipple and skin sparing procedures. Nipple-sparing mastectomy (NSM) with reconstruction technology offers the opportunity to preserve the shape of both the breast and the nipple-areola complex.

This study will evaluate the safety and effectiveness of the da Vinci Surgical Systems in NSM procedures.

ELIGIBILITY:
Inclusion Criteria:

* Female between ages 18-80.
* BMI ≤ 29.
* Candidate for an NSM procedure.
* At increased risk for breast cancer and is seeking prophylactic NSM surgery or subject has breast cancer in one breast and is seeking prophylactic NSM on contralateral side.
* Breast ptosis ≤ Grade 2.
* Cup size ≤ C.
* No presence of occult cancer on the side for which she is seeking prophylactic NSM surgery as confirmed by physical exam and by preoperative imaging per institution's guidelines.

Exclusion Criteria:

* Current or prior history of ipsilateral in-situ or invasive breast carcinoma on the breast for which she is seeking prophylactic NSM surgery.
* Previous breast surgery of the ipsilateral breast (excluding needle or core biopsies and excisional biopsies performed more than 1 year prior).
* Current history of smoking or has smoked within 1 year of screening.
* Skin conditions
* Uncontrolled diabetes mellitus.
* Previous chemotherapy or radiation
* High risk for anesthesia or significant medical comorbidities
* Contraindicated for general anesthesia or surgery.
* Known bleeding or clotting disorder.
* Pregnant or suspected to be pregnant or is lactating.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2021-03-26 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness: No conversions to open NSM | Assessed during surgery
  Conversion is defined as conversion of da Vinci robotic-assisted surgery to open surgery
Primary Safety: Incidence of adverse events | Assessed during surgery to 42 days after surgery
  Incidence of intraoperative and post-operative procedure and device-related adverse events

OTHER OUTCOMES:
Incidence of breast cancer | Annual through 5 year post-operatively
  Occurrence and recurrence of breast cancer
Patient reported outcomes | Pre-operatively, post-operatively at 42 days, annually through 5 years
  BREAST-Q
Long-term safety: incidence of adverse events | Annually through 5 years post-operatively
  Incidence of breast procedure-related adverse events during long-term follow up

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Mayo Clinic Florida, Jacksonville, Florida
  - NorthShore University Health System, Evanston, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Northwell Health, New Hyde Park, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No